CLINICAL TRIAL: NCT03370731
Title: The Impact of Adenotonsillectomy Versus Nonsurgical Management on Quality of Life for Children With Controversial Diagnoses of Obstructive Sleep Apnea Under Different Criteria
Brief Title: Surgical Versus Nonsurgical Treatment on Quality of Life for Children With Controversial OSA Diagnoses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: Beijing Children's Hospital (Other); Shanghai 6th People's Hospital (Other); Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRECKY2017-032-1
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Obstructive Sleep Apnea of Child
Keywords: pediatric; obstructive sleep apnea; polysomnography; quality of life; adenotonsillectomy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adenotonsillectomy (Experimental): Surgical management, i.e. adenotonsillectomy, including adenoidectomy, tonsillectomy or adenoidectomy combined tonsillectomy
  Interventions: Procedure: adenotonsillectomy
- Nonsurgical management (Other): Nonsurgical management, including nasal irrigation, inhaled corticosteroids etc.
  Interventions: Other: Nonsurgical management

INTERVENTIONS:
Procedure: adenotonsillectomy — Resection of adenoidal tissue or hypertrophy tonsils by radiofrequency ablation or other methods.
  Arms: Adenotonsillectomy
Other: Nonsurgical management — Nasal Irrigation or inhaled corticosteroids, etc.
  Arms: Nonsurgical management

SUMMARY:
Obstructive sleep apnea (OSA) is a disease characterized by repeated partial or complete upper airway collapse during sleep, accompanied by arousals or oxygen desaturation. It was reported to affect 5.7 %~9.6 % of pediatric population in western countries and 5.5 %~7.8 % in China. Children's physical developing and brain functioning as well as quality of life (QoL) could be greatly impaired if the disease was left untreated.

Polysomnography (PSG) was recognized as gold standard for diagnosing OSA. However, for pediatric OSA, there exists dispute on the PSG diagnostic criteria.

Pediatric OSA was mostly caused by hypertrophy of adenoid or palatine tonsillar. For those PSG validated patients, nonsurgical management was often prescribed, in addition, surgical intervention, i.e. adenotonsillectomy was also commonly applied and had been proved efficient both in terms of PSG and in terms of symptoms, behaviors and QoL rated by caregivers. However, for children with controversial diagnoses by ATS and ICSD-3, little was known about whether surgical or nonsurgical management was effective.

We aim at investigating the effect of adenotonsillectomy versus nonsurgical management on QoL in these subjects. And the hypothesis is that adenotonsillectomy improves QoL better than nonsurgical management in children with controversial diagnoses of OSA by ATS and ICSD-3.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a disease characterized by repeated partial or complete upper airway collapse during sleep, accompanied by arousals or oxygen desaturation. It was reported to affect 5.7 %~9.6 % of pediatric population in western countries and 5.5 %~7.8 % in China. Children's physical developing and brain functioning as well as quality of life (QoL) could be greatly impaired if the disease was left untreated.

Polysomnography (PSG) was recognized as gold standard for diagnosing OSA. However, for pediatric OSA, there exists dispute on the PSG diagnostic criteria. The American Thoracic Society standard (ATS) treated children with AHI > 5/H or obstructive apnea index (OAI) > 1/H as abnormal, while the International Classification of Sleep Disorder standard (ICSD-3) used obstructive apnea-hypopnea index (OAHI) ≥ 1/H. Due to the differences of the above criteria, there were a set of children whose diagnoses were controversial, making the treatment decision rather thorny.

Pediatric OSA was mostly caused by hypertrophy of adenoid or palatine tonsillar. For those PSG validated patients, nonsurgical management was often prescribed, in addition, surgical intervention, i.e. adenotonsillectomy was also commonly applied and had been proved efficient both in terms of PSG and in terms of symptoms, behaviors and QoL rated by caregivers. However, for children with controversial diagnoses by ATS and ICSD-3, little was known about whether surgical or nonsurgical management was effective.

We aim at investigating the effect of adenotonsillectomy versus nonsurgical management on QoL in these subjects. And the hypothesis is that adenotonsillectomy improves QoL better than nonsurgical management in children with controversial diagnoses of OSA by ATS and ICSD-3.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 2 to 14 years
* Complaints of habitual sleep snoring, apnea, mouth breathing, daytime somnolence
* ATS positive (AHI > 5/H or OAI > 1/H) & ICSD-3 negative (OAHI < 1/H) or ATS negative (AHI ≤5 /H or OAI ≤ 1/H) & ICSD-3 positive (OAHI ≥ 1/H)

Exclusion Criteria:

* Aged below 2 or above 14 years
* Unconscious
* Facial dysplasia
* Neuro-psychological diseases
* Having taken spirit or nervous system drugs within 3 months
* Diagnosed with acromegaly, hypothyroidism, vocal cord paralysis, laryngeal spasm, epilepsy， narcolepsy or neuromuscular disease
* Having received systematic treatment for OSA (having used a ventilator for more than 1 month, or having received adenotonsillectomy.)
* Caregivers did not fill out the questionnaire either pre or postoperatively

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
OSA-18 | At least 6 month.
  A quality of life questionnaire OSA-18 was used. It was presented by Franco RA and colleagues, and proven good test-retest reliability and internal consistency and widely used for evaluating QoL of snoring children. In this study, QoL was assessed by OSA-18. It was filled by the caregivers with the assistance of designated medical staff before PSG monitoring as well as when subjects were followed up. The questionnaire consisted of 18 items and 5 domains: sleep disturbance, physical symptoms, emotional symptoms, daytime function, and caregiver concerns. Each item was scored 1 to 7, and the total score ranged from 18 to 126 (the higher the score, the more severe the situation).

CONTACTS AND LOCATIONS:
Overall Officials: Demin Han, Prof., Study Director — Beijing Tongren Hospital
Locations (4):
- China (4):
  - Beijing Children's Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Beijing, Beijing Municipality
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Shanghai 6th People Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Garetz SL, Mitchell RB, Parker PD, Moore RH, Rosen CL, Giordani B, Muzumdar H, Paruthi S, Elden L, Willging P, Beebe DW, Marcus CL, Chervin RD, Redline S. Quality of life and obstructive sleep apnea symptoms after pediatric adenotonsillectomy. Pediatrics. 2015 Feb;135(2):e477-86. doi: 10.1542/peds.2014-0620. Epub 2015 Jan 19. PMID 25601979
- [Result] Franco RA Jr, Rosenfeld RM, Rao M. First place--resident clinical science award 1999. Quality of life for children with obstructive sleep apnea. Otolaryngol Head Neck Surg. 2000 Jul;123(1 Pt 1):9-16. doi: 10.1067/mhn.2000.105254. PMID 10889473
- [Result] Baldassari CM, Mitchell RB, Schubert C, Rudnick EF. Pediatric obstructive sleep apnea and quality of life: a meta-analysis. Otolaryngol Head Neck Surg. 2008 Mar;138(3):265-273. doi: 10.1016/j.otohns.2007.11.003. PMID 18312869
- [Result] Venekamp RP, Hearne BJ, Chandrasekharan D, Blackshaw H, Lim J, Schilder AG. Tonsillectomy or adenotonsillectomy versus non-surgical management for obstructive sleep-disordered breathing in children. Cochrane Database Syst Rev. 2015 Oct 14;2015(10):CD011165. doi: 10.1002/14651858.CD011165.pub2. PMID 26465274
- [Result] Mandavia R, Dhar V, Kapoor K, Rachmanidou A. Quality of life assessment following adenotonsillectomy for obstructive sleep apnoea in children under three years of age. J Laryngol Otol. 2012 Dec;126(12):1241-6. doi: 10.1017/S002221511200237X. Epub 2012 Oct 30. PMID 23110961